CLINICAL TRIAL: NCT02695849
Title: An Epidemiology Study of the Prevalence of Epidermal Growth Factor Receptor (EGFR) Mutations in Patients Diagnosed With Non-squamous Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Prevalence of EGFR Mutations in Participants With NSCLC
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25269
Record Dates: First submitted 2016-02-25; First posted 2016-03-01 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-small cell lung cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- NSCLC Participants: Participants with non-squamous NSCLC will be enrolled in this study.

SUMMARY:
This is a non-interventional, local, multicenter, cross-sectional study to determine the prevalence of epidermal growth factor receptor (EGFR) mutations in participants diagnosed with non-squamous non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signature
* Jordanian male and female participants greater than or equal to (>=) 18 years of age
* Histologically confirmed NSCLC
* Not participating in a study that involves an investigational agent within 30 days prior to enrollment

Exclusion Criteria:

* Other primary malignancy
* Fine needle aspiration samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with non-squamous non-small cell lung cancer (NSCLC)
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2012-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with EGFR mutations | Day 1

SECONDARY OUTCOMES:
Percentage of Participants with types of EGFR mutations | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Amman, Jordan